CLINICAL TRIAL: NCT04343300
Title: The Effectiviness of Pilates on the Risk of Fall in Healthy Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Larissa Donatoni da Silva, Principal investigator, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LdaSilva; CAPES (Other Grant/Funding Number: Coordenação de Aperfeiçoamento de Pessoal de Nivel Superior)
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-04

CONDITIONS: Healthy
MeSH Terms: interventions — Exercise Movement Techniques; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No

ARMS (2):
- Control group (Other): Control group without Pilates exercise during 12 weeks Participants were advised to keep their routine Falls diary calendar
  Interventions: Other: exercise without Pilates
- Pilates group (Experimental): Pilates classes were held twice weekly for one hour. The classes were divided into a warm-up, mat Pilates with accessories and a cool-down. Participants used small items of equipment such as bands, circles or rings, blocks, spyke balls and foam rollers. The intervention lasted 12 weeks; the classes were supervised twice a week. The supervised exercises were evaluated every four weeks (frequency and intensity) focused on the lower limb (muscles related to gait), core and trunk (muscles related to posture). The participants were asked to perform supplementary at-home workouts three times a week using a booklet and video that was provided to the participants. The video and booklet to introduce the six principles of Pilates, warm-up exercises, exercises on the chair, mat Pilates exercises and cool-down exercises. Participants were advised to perform these exercises three times a week for 30 minutes at home.
  Interventions: Other: Pilates

INTERVENTIONS:
Other: Pilates — Intervention of12 weeks of Pilates
  Arms: Pilates group
Other: exercise without Pilates — exercise without Pilates
  Arms: Control group

SUMMARY:
This research examine the effectiveness of a Pilates intervention for reducing the risk of falls among adults aged over 65 years. The effects were measured the Pilates classes with a supplementary home-based exercises in two phases: Phase I investigated (Mat Pilates supervised with a supplementary home-based Pilates exercise for the pre and post-test of 6 weeks intervention. Eligible 32 participants). The main study randomised controlled trial (phase II) investigate whether a Pilates intervention of 12 weeks with a supplementary at home program is effective in reducing falls risk factors. Pilates group which practiced Pilates and the control group which did not practice Pilates The aim of the study is to identify whether spatiotemporal gait parameters, mobility, postural stability parameters of anteroposterior and mediolateral (AP-ML), functional mobility, fear of falling and physical activity changes.

DETAILED DESCRIPTION:
There are a lack of studies evaluating the spatiotemporal parameters of gait, fear of falling, and physicial activity after a Pilates intervention. The inclusion criteria were healthy older adults (≥ 65 years). Demographic details: age, gender, height, weight, Body Mass Index, health status, 2 question of fear and previous falls (one year). Screening test: The Montreal cognitive MOCA test. Participants were assessed using the following fall-predictor measures. Primary outcomes: the 16-item Falls Efficacy Scale-International (FES-16), and the Footwork Pro pressure plate system. Secondary outcomes: the Timed Up and Go (TUG), the GAITRite system, the International Physical Activity Questionnaire (IPAQ), the Functional Reach Test (FRT). The randomised controlled trial, eligible n=61 participants and randomise allocated into control group (no exercise) and Pilates group. The Pilates intervention took place at the Aras Moyola building, NUI Galway.The instructor is fully qualified to carry out the Pilates programme. The instructor is a qualified physiotherapist and has undertaken courses clinical Pilates in Valeria Figueireido International and Body Control Pilates for older adults. The video and booklet were built by the PI. The booklet contains pictures demonstrated by the instructor. Participants also had access to the home-based Pilates exercise video via a Dropbox link sent to their email by PI. The instructor demonstrated, explained and showed the exercises through the video to the participants during the first supervised Pilates class which participants also performed the home-based exercises. Feedback notes and comments were also taken from the participants. The participants were asked to give feedback on the same day as the assessments (Post-test). Questionnaire of Pilates exercises applied for the participants after Pilates 24 sessions supervised completed and a diary calendar of falls during the period of the intervention of 12 weeks, phone calls and e-mails were provided by the PI.

ELIGIBILITY:
Inclusion Criteria:

Those over 65 years older, both male and female, healthy and able to attend the Pilates sessions regularly were included. Those included had not had surgery in the past six months, had no restriction recommended by their General Practitioner and had a Montreal Cognitive Assessment score of over 26

Exclusion Criteria:

Those excluded had a MOCA score of less than 26, had a fall in the last six months. had several pain, had acute inflammation, had a history of neurological illness, had medical and pharmacologic contraindications to exercise, vertigo or had a strong exercise routine already.

Ages: 65 Years to 87 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Falls Efficacy Scale | up to 12 weeks
  Participants should answer items thinking about how they usually do the activity and they should answer items to show how concerned they would be about falling: 1 = not at all concerned 2 = somewhat concerned 3 = fairly concerned 4 = very concerned. Total score ranging from 16 (not at all) to 64 (very much).
Platform Footworkpro Pressure plate | up to 12 weeks
  Measure the two parameters of stabilometry in mediolateral (cm) and anteroposterior (cm) sway in static position performance

SECONDARY OUTCOMES:
Functional Reach Test (FRT) | Baseline, post-test 12 weeks
  Mobility and balance
Functional Reach Test (FRT) | Baseline, post-test 6 weeks
  Mobility and balance
Timed Up and Go (TUG) | Baseline, post-test 12 weeks
  Functional mobility
Timed Up and Go (TUG) | Baseline, post-test 6 weeks
  Functional mobility
GAITRite® system | Baseline, post-test 12 weeks
  Spatial and temporal parameters of gait
GAITRite® system | Baseline, post-test 6 weeks
  Spatial and temporal parameters of gait
The short International Physical Activity Questionnaire | Baseline, post-test 12 weeks
  Measure daily physical activity such as leisure time, domestic and gardening (yard) activities, work-related and transport-related activities. The total scores of walking; moderate, and vigorous-intensity activity described the overall level of activity in (METs) metabolic equivalent minutes per week, calculates as the MET intensity multiplied per min for each activity during the last seven days such as walking=3.3 METs, Moderate PA= 4.0 METs and Vigorous PA= 8.0 METs. The total MET min/week = (walk MET*min*days) + (Mod MET*min*days) +Vig METs*min*days) (http://www.ipaq.ki.se).
The short International Physical Activity Questionnaire | Baseline, post-test 6 weeks
  Measure daily physical activity such as leisure time, domestic and gardening (yard) activities, work-related and transport-related activities. The total scores of walking; moderate, and vigorous-intensity activity described the overall level of activity in (METs) metabolic equivalent minutes per week, calculates as the MET intensity multiplied per min for each activity during the last seven days such as walking=3.3 METs, Moderate PA= 4.0 METs and Vigorous PA= 8.0 METs. The total MET min/week = (walk MET*min*days) + (Mod MET*min*days) +Vig METs*min*days) (http://www.ipaq.ki.se).

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Donatoni da Silva, Phd student, Principal Investigator — National University of Ireland, Galway

IPD SHARING:
Plan to Share IPD: Undecided
check